CLINICAL TRIAL: NCT01999387
Title: Follow up of Patients After Oral Immunotherapy for Cow's Milk, Eggs and Peanuts
Acronym: OIT followup
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 41/13
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-06

CONDITIONS: Allergy
Keywords: food; consumption
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood tests
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Completed OIT: Patients who completed OIT >6 months prior to enrollment
  Interventions: Dietary Supplement: Allergenic food

INTERVENTIONS:
Dietary Supplement: Allergenic food

SUMMARY:
Food allergy is a potentially life threatening condition. The current practice consists of elimination diet and injectable epinephrine in case of a reaction.

Recently, oral immunotherapy has emerged as a treatment for food allergy in milk eggs and peanuts.

We conduct an oral immunotherapy program with ~500 patients so far. In this study we intent to follow patients who completed the program and assess their allergy status and quality of life.

DETAILED DESCRIPTION:
Food allergy is a potentially life threatening condition. The current practice consists of elimination diet and injectable epinephrine in case of a reaction.

Recently, oral immunotherapy (OIT) has emerged as an treatment for food allergy in milk eggs and peanuts. Since 4/2010,a clinical OIT program for milk eggs and peanuts is performed at the Institute fir Allergy Asthma and Immunology at Assaf Harofeh Medical Center with ~500 patients so far. Patients with IgE-mediated food allergy that are >4 years old are eligible.

In this study we intent to follow patients who completed the program. Patients will fill a questionnaire regarding current consumption of the allergenic food, adverse reactions experienced and treatments required including the use of EpiPen. Patients underwent skim prick tests (SPT) for the allergenic food prior to initiation and treatment and will undergo SPT again upon entering the study. Blood tests for IgE, IGG4, basophil activation and cytokines will be obtained.

Patients who are not consuming the allergenic food regularly will undergo an oral food challenge in clinic.

ELIGIBILITY:
Inclusion Criteria:

* age>4 years old IgE mediated allergy to milk eggs or peanuts Completion of OIT >6 months ago

Exclusion Criteria:

* Non approval to participate

Ages: 4 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients > 4 years old with IgE mediated allergy to cow;s milk, eggs or peanuts who completed an OIT program >6 months ago
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Allergenic food consumption questionnaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yitzhak Katz, MD, Principal Investigator — Asaf Harofeh Medical enter
Locations (1):
- Asaf Harofeh Medical Center, Ẕerifin, Israel, Israel